CLINICAL TRIAL: NCT00572923
Title: Concurrent Chemo-Radiotherapy for Limited Disease Small Cell Lung Cancer (LD-SCLC) on Basis of FDG-PET-Scans
Acronym: BRONC 45 15
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: MAASTRO clinic, MAASTRO clinic
Other Study IDs: BRONC 45, 1.5
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Small Cell Lung Cancer
Keywords: radiotherapy; LD-SCLC; stage I-III small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Inclusion criteria
  * Histological or cytological proven SCLC
  * UICC stage I-III, "limited disease"
  * Performance status 0-2
  * FeV1 and DLCO at least 30% of age-predicted value
  Exclusion criteria:
  * Not SCLC or mixed SCLC and other histologies (e.g. non-small cell carcinoma)
  * stage IV
  * performance status 3 or more
  * FeV 1 or DLCO< 30% of the age-predicted value

SUMMARY:
Our group has shown that the omission of elective nodal irradiation on the basis of CT scans in patients with LD-SCLC lead to a higher than expected isolated nodal recurrence in the ipsilateral supraclavicular area. We have previously also shown that selective mediastinal nodal radiation on basis of FDG-PET scans in NSCLC is safe and reduces the radiation fields and hence toxicity. As the accuracy of FDG-PET scans is also in SCLC higher than CT, we will investigate the safety of selective nodal irradiation in LD-SCLC patients treated with concurrent chemo-radiation.

DETAILED DESCRIPTION:
Eligible patients (see below) will receive radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes on FDG-PET scan to a dose of 45 Gy in 30 fractions in 3 weeks (1.5 Gy BID with minimum 6 h interfraction interval).

Dose-constraints: MLD > 20 Gy. In that case, CT-based replanning will be done after 1 week of treatment and shrinking field techniques will be used if appropriate.

The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic.

Radiotherapy shall start during the first cycle of carboplatin and etoposide chemotherapy.

Chemotherapy (standard schedule in the Comprehensive Cancer Centre Limburg region):

* carboplatin AUC 5 day 1
* etoposide 120 mg/m2 days 1-3

Q 3 weeks; 5 cycles

In patients with no progression and a WHO PS 0-2, after the completion of chemotherapy, PCI will be given (25 Gy in 10 fractions, QD)

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven SCLC
* UICC stage I-III, "limited disease"
* Performance status 0-2
* FeV 1 and DLCO at least 30% of the age-predicted value

Exclusion Criteria:

* Not SCLC or mixed SCLC and other histologies (e.g. non-small cell lung carcinoma)
* UICC stage IV
* Performance status 3 or more
* FeV 1 and DLCO < 30% of the age-predicted value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Histological or cytological proven SCLC
  * UICC stage I-III, "limited disease"
  * Performance status 0-2
  * FeV 1 and DLCO at least 30% of the age-predicted value
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2006-08; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
isolated Nodal Recurrences | 18 months post-treatment

SECONDARY OUTCOMES:
overall survival | 18 months post-treatment
progression-free interval | 18 months post-treatment
dyspnea (CTCAE 3.0) | 18 months post-treatment
dysphagia (CTCAE 3.0) | 18 months post-treatment
patterns of recurrence | 18 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD,PhD, Principal Investigator — MAASTRO clinic, Maastricht Radiation Oncology
Locations (1):
- MAASTRO clinic, Maastricht Radiation Oncology, Maastricht, Netherlands